CLINICAL TRIAL: NCT00316446
Title: A Prospective Double Blind Pilot Study to Determine the Incidence of Postoperative Hypoventilation in Patients With Clinically Significant Obesity Who Have Undergone Gastric Bypass Procedures Under General Anesthesia
Brief Title: Study to Determine Incidence of Hypoventilation in Patients Who Have Undergone Gastric Bypass
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: USF1
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Morbid Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if gastric bypass patients experience hypoventilation in the immediate postoperative period, and to what degree.

DETAILED DESCRIPTION:
We propose to determine if patients with clinically significant obesity (body mass index, BMI, between 40 kg/m2 and 85 kg/m2), who have undergone gastric bypass procedures under general anesthesia hypoventilate during the initial twenty-four hour postoperative period, and if so, to what degree. Adequacy of ventilation will be assessed by serial arterial blood analyses. Patients will be monitored for SpO2 in the preoperative holding area, in the operating room, and the post-anesthesia care unit (PACU) by conventional and study pulse oximeters. SpO2 data will be collected continuously and recorded on the study pulse oximeter for the entire study period. Arterial blood samples will be drawn for analysis every four hours by in-dwelling arterial catheter, using standard sterile technique. Hypoventilation is defined as an increase in PaCO2 five or more mm Hg above patient's baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 65 years of age
* Clinically significant obesity with a BMI between 40 and 85
* Candidates approved for gastric bypass surgery at Tampa General Hospital (*Please note: authorization for gastric bypass will be completed prior to enrollment in study; this study does not pay for the cost of the operation.)
* American Society of Anesthesiologists (ASA) Physical Status Classification I-III
* Able to understand and sign informed consent

Exclusion Criteria:

* Patients not able to understand the informed consent process, or unable to understand the research protocol
* Patients in which placing an arterial catheter would pose a clinically unacceptable health risk, e.g., bleeding disorders, radial artery malformation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female adult patients (age 18-65) with clinically significant obesity (body mass index (BMI) between 40-85 kg/m2), who are approved for gastric bypass surgery for weight loss. Patients must have documented obstructive sleep apnea and use continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP), and have an American Society of Anesthesiologists (ASA) Physical Status Classification I-III.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott F Gallagher, MD, Principal Investigator — University of South Florida, Department of Surgery
Locations (1):
- University of South Florida, Department of Surgery at Tampa General Hospital, Tampa, Florida, United States